CLINICAL TRIAL: NCT01067209
Title: Reversal of Obesity- and Diabetes-related Cardiomyopathy in Patients Who Have Undergone Gastric Bypass Surgery.
Brief Title: Reversal of Obese/Diabetic Cardiomyopathy After Gastric Bypass Surgery
Acronym: DRTC
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 09-1295
Record Dates: First submitted 2010-02-09; First posted 2010-02-11 (Estimated); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Cardiomyopathy
Keywords: Reversal of Obesity-related and Diabetic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathies; Diabetic Cardiomyopathies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Diabetic/Obese Gastric bypass patients: Subjects with obesity including those with known diabetes or those with a high likelihood of diabetes who will undergo gastric bypass surgery.

SUMMARY:
The overall purpose of this study is to evaluate the effect of gastric bypass surgery-induced weight loss on the heart's function and on fat deposits in the heart muscle.

DETAILED DESCRIPTION:
Diabetes is a major risk factor for heart failure. Moreover, patients with diabetes and heart failure have a worse survival than those without diabetes. We know that patients with diabetes have altered heart metabolism, structure, and function. It is unclear if these alterations can be ameliorated with weight loss. We would like to learn whether cardiac metabolism, structure, and function in diabetic patients with heart failure symptoms can be improved with marked weight loss after gastric bypass surgery.

Study Day 1. Screening. We will screen subjects with known diabetes or those with a high likelihood of diabetes who will undergo gastric bypass surgery. We will approach all patients at the Bariatric Surgery clinic regarding enrollment in our study. If they agree to participate, they will answer simple questionnaires re: medical history, obesity information, and MRI/MRS exclusion (see Appendices). We will obtain their permission to review their medical charts.

Study Day 2. Screening will include a physical examination and phlebotomy for a complete blood count, oral glucose tolerance test, & comprehensive metabolic profile and a screening rest and stress echocardiogram. The rest and stress echocardiogram will be used to exclude cardiac abnormalities other than diastolic dysfunction. Optison™ or Definity will be used as needed for the echocardiograms. We will determine the subjects' fat and fat-free mass using dual-energy X-ray absorptiometry (DXA) imaging at the Center for Applied Research Sciences unit.

Study Day 3. Baseline Imaging Studies. Subject preparation. We expect 30 subjects to complete our study's screening tests and meet our study criteria. The evening before imaging Study Days 3 & 4, subjects will be admitted to The Center for Applied Research Sciences Intensive Research Unit in order to standardize their metabolic milieu for their myocardial fat imaging studies. At 1800, subjects will ingest a standard meal containing a total of ~700 kcal for the subjects. Carbohydrate, fat, and protein will represent 55, 30, and 15%, respectively, of total energy intake. At 2000, subjects will ingest a defined liquid formula snack containing 250 kcal, 40 g carbohydrate, 6.1 g fat, and 8.8 g protein (Ensure, Ross Laboratories, Columbus, OH). After this snack, all subjects will fast until completion of the study the following day. Subjects will be given a lunch after completing their imaging studies. Magnetic resonance imaging (MRI). Subjects will be placed in the gantry of the scanner. Examinations will be performed on the 1.5T scanner using ECG gating, breath-hold, and a chest array coil This same scanner will be used for 1H-Magnetic resonance spectroscopy (MRS). The MRS protocol is based on a free-breathing, point-resolved spectroscopy (PRESS) sequence with both ECG and two-dimensional respiratory gating optimized for accuracy and robustness. Subject care. All subjects will be given a lunch, prepared at the Intensive Research Unit after imaging is completed. All imaging should be completed by 12PM. If the physician monitoring the subject determines that the subject would benefit from furosemide 20mg, p.o. x 1, or KCl, p.o. - a 10 day course may be provided (with a follow-up K+ check). Patients' physicians would be notified of any changes. We request subjects stay on their same medical regimen throughout the testing period. We recognize that this may not be possible for all subjects.

Gastric bypass. Subjects will undergo surgery after Study Day 3. The same surgeon (J.C.E.) will perform all bypass procedures using standard techniques. Briefly, a small (~20 mL) proximal gastric pouch will be created by stapling across the stomach, and a 150 cm Roux-Y limb constructed by transecting the jejunum 30cm distal to the ligament of Treitz and creating a jejunojejunostomy 150 cm distal to the transection.

Study Day 4. Imaging Studies - 3 months after surgery. Subjects will undergo the same imaging studies under the same conditions and in the same order as on Study Day 3 except that subjects on Day 4 will also undergo a resting echocardiogram for diastolic function.

ELIGIBILITY:
Inclusion Criteria:

* All subjects will have type 2 diabetes or be at risk for type 2 diabetes and have a BMI>30kg/m2.
* Subjects must be between the ages of 35 and 70 years, in order to limit the confounding affect of age on our endpoints.
* 23 Subjects must also meet the following definition of diastolic dysfunction:

  * 1) meet Framingham criteria for heart failure (see Appendix),
  * 2) have an ejection fraction >45% based on the rest portion of the screening echocardiography,
* 24 To determine if potential subjects meet these criteria, they will

  * 1) be interviewed,
  * 2) their clinical charts reviewed, by the research study coordinator and/or the PI, and
  * 3) undergo a history and physical by the PI (Study Day 2) and undergo screening studies.

Exclusion Criteria:

* Subjects who are <35 or >70 years,
* current smokers, not obese,
* unstable,
* not able to lie flat for the imaging studies,
* not ambulatory,
* unable to give informed consent,
* pregnant, lactating will be excluded.
* Those who have a condition that may masquerade as diastolic heart failure (e.g. constrictive pericarditis) will be excluded based on the screening echocardiogram;
* those who have atrial flutter or fibrillation,
* evidence of other major systemic diseases (e.g., cancer),
* an ejection fraction <45%, >class I hypertension or who are taking more than 1 medication (other than a diuretic) for hypertension will be excluded.
* We will not exclude patients with sleep apnea because data suggest it does not affect left ventricular (LV) diastolic function, but we will ask about it on a questionnaire for better phenotyping of the subjects.25
* We will exclude patients with significant pulmonary hypertension (peak artery pressure>55mmHg), since most patients with diastolic dysfunction have a pressure lower than this, and a pressure greater than this may indicate other cardiopulmonary pathology.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese patients +/- known diabetes who will undergo gastric bypass surgery.
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2010-01; Primary Completion 2013-02-14 (Actual); Study Completion 2013-02-14 (Actual)

PRIMARY OUTCOMES:
Primary outcome measure: cardiac function, myocardial fat deposition | the time frame of the study

SECONDARY OUTCOMES:
Plasma lipidomics, liver fat deposition | the time frame of the study

CONTACTS AND LOCATIONS:
Overall Officials: Linda R Peterson, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States